CLINICAL TRIAL: NCT00288431
Title: A Phase 1B, Sequential Cohort, Dose Escalation Trial to Determine the Safety, Tolerability and Maximum Tolerated Dose of Oral AP23573 in Combination With Doxorubicin
Brief Title: Safety, Tolerability and Maximum Tolerated Dose of Oral AP23573 in Combination With Doxorubicin (8669-015)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-015; AP23573-05-107
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Cancer; Sarcoma
Keywords: cancer; sarcoma
MeSH Terms: conditions — Neoplasms; Sarcoma | interventions — ridaforolimus; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Different schedules and routes of administration of AP23573 will be examined. For each schedule, AP23573 + Doxorubicin will be co-administered on Day 1 of a 3-week cycle. AP23573 will be given orally and will range in dose from 10-30 mg per dose.
  Interventions: Drug: ridaforolimus; Drug: Doxorubicin

INTERVENTIONS:
Drug: ridaforolimus — Different schedules and routes of administration of AP23573 will be examined. For each schedule, AP23573 + Doxorubicin will be co-administered on Day 1 of a 3-week cycle. AP23573 will be given orally and will range in dose from 10-30 mg per dose.
  Other Names: deforolimus; AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009
Drug: Doxorubicin — administered at 60 mg/m2 intravenously every 3 weeks

SUMMARY:
This study is designed to determine the safety, tolerability and maximum tolerated dose of Oral AP23573 in combination with Doxorubicin

DETAILED DESCRIPTION:
The primary objective is to determine the maximum tolerated dose (MTD) of AP23573 in combination with doxorubicin, to characterize the safety profile of AP23573 in combination with doxorubicin, and to examine the pharmacokinetics of AP23573 and doxorubicin when given in combination to patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with a histological/cytological diagnosis of advanced tumor, preferentially breast, sarcoma, ovarian, endometrial or other tumor types for which treatment with anthracycline therapy is indicated
* Prior cumulative doxorubicin exposure less than 400 mg/m2
* An ECOG performance status of 0 or 1
* Adequate cardiovascular function
* Measurable disease according to modified RECIST criteria
* Adequate hematological, renal and hepatic functions
* Able to understand and give voluntary written informed consent

Exclusion Criteria:

* Women who are pregnant or lactating
* Presence of active brain metastases. Patients with treated brain metastases will be eligible if they are on a stable dose of corticosteroids or are without change in brain disease status for at least 4 weeks following related therapy (e.g., whole brain radiation, surgery)
* Prior treatment with CCI-779, rapamycin, or any other mTOR inhibitor
* Prior anticancer treatment (chemotherapy, radiotherapy, hormonal, immunotherapy, biological response modifiers, signal transduction inhibitors, etc) within 4 weeks prior to the first dose of AP23573; the interval is ≥ 2 weeks for signal transduction inhibitors with a half-life known to be <24 hours, and is ≥ 6 weeks for nitrosourea or mitomycin. Exception: Concurrent treatment with LHRH agonists is allowed for patients with prostate cancer.
* Ongoing toxicity associated with prior anticancer therapy other than alopecia and ≤ Grade 1 peripheral neuropathy by NCI toxicity criteria
* Another primary malignancy within the past three years (except for non-melanoma skin cancer and cervical carcinoma in situ)
* Known or suspected hypersensitivity to any excipient contained in the study drug
* Known Grade 3 or 4 hypersensitivity to macrolide antibiotics (e.g., clarithromycin, erythromycin, azithromycin)
* Significant uncontrolled cardiovascular disease
* Any active infection requiring prescribed intervention
* Any other concurrent illness which, in the opinion of the investigator, would either compromise the patient's safety or interfere with the evaluation of the safety of the study drug
* Any pre-existing malabsorption syndrome, irritable bowel syndrome or other clinical situation which could affect oral absorption
* Concurrent treatment with immunosuppressive agents other than prescribed corticosteroids at stable doses for ≥ 2 weeks prior to first planned dose of study drug
* Concurrent treatment with medications that induce or inhibit cytochrome P450 (CYP3A)
* Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within 2 weeks prior to the first dose of AP23573

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
determine the maximum tolerated dose (MTD) of oral AP23573 in combination with doxorubicin | Duration of study

SECONDARY OUTCOMES:
Describe the antitumor activity of the study drug combination for each dosing schedule | Duration of study
examine the pharmacokinetics of oral AP23573 and doxorubicin when given in combination | Duration of study
Examine pharmacodynamic characteristics of AP23573 for those patients enrolled into the expanded MTD cohorts only | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC